CLINICAL TRIAL: NCT04601727
Title: Oral & Faecal Microbiota Analysis in Patients With Rectal Cancer Requiring Pre-operative Therapy Before Surgery, & Correlation With Response. (The MicrobRect Study).
Brief Title: Oral & Faecal Microbiota Analysis in Patients With Rectal Cancer Requiring Pre-operative Therapy Before Surgery, & Correlation With Response
Acronym: MICROBRECT
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-014-20
Record Dates: First submitted 2020-09-21; First posted 2020-10-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 16srRNA analysis of faeces and saliva before and after neoadjuvant chemoradiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal cancer patients
  Interventions: Diagnostic Test: 16srRNA pyrosequencing analysis of microbiota of saliva and faeces

INTERVENTIONS:
Diagnostic Test: 16srRNA pyrosequencing analysis of microbiota of saliva and faeces — No intervention in this study

SUMMARY:
Rectal cancer is a common pathology which is treated by a multimodal approach. Those tumours in the rectum that are locally advanced are treated with neoadjuvant chemoradiotherapy before an operation. This aims to reduce the size of the tumour and increase the change of a complete resection. The degree of shrinkage of a rectal cancer to pre-operative treatment is influenced by the immune system. In some other cancers there is evidence that the bacteria living in our mouth & in the large bowel influence the way the body responds a cancer. In this study patients with rectal cancer requiring radiotherapy before surgery will be asked to give samples of saliva & bowel motions before chemoradiotherapy & again before surgery. These samples will have the type and number of bacteria analysed, as well as levels of key metabolic products of these bacteria. The results will be compared with the response, as assessed by the pathologist using standard criteria, of the rectal to the radiotherapy.

DETAILED DESCRIPTION:
Introduction:

Pelvic radiotherapy (VMAT) and chemotherapy are used in margin threatened rectal cancer to reduce the cancer and achieve a clear circumferential resection margin (CRM), facilitating potentially curative surgery. In 15 to 20% of cases, the pre-operative chemoradiotherapy potentially completely treats the cancer raising the possibility to avoid surgery altogether. Increasing the number of patients who are able to be cured without surgery is a research priority for the NCRI Colorectal Studies Group in UK. Other patients have some reduction in the size of the malignancy (a partial response) and others have a minimal response to the pre-operative therapy. As yet, it remains unclear as to the mechanism of response of the cancer to neoadjuvant therapy.

Understanding what biological factors influence response is important in order to improve the outcomes in rectal cancer. There is evidence that the innate immune system has a role in the degree of response. An increased degree of response (as measured by tumour regression grading) is associated with an increased abundance of natural killer (NK) CD56+ve cells. In mouse models the gut microbiome can modulate the tumour-immune microenvironment and T cell responses in colonic cancer. In addition some bacteria that are associated with colorectal cancer, such as F. nucleatum, are indigenous to the human oral cavity, and evidence that patients with colorectal cancer have a distinctive oral microbiota.

Clinical studies are needed to investigate the role of the oral & faecal microbiome in response to pre-operative treatment. If there is evidence of an association, the challenge will then be to explore if this can be modulated to increase response. Alternatively, the pre treatment microbiota profile may be able to be used as a predictor of response to neoadjuvant therapy.

This is a pilot study to assess the feasibility and acceptability to patients in providing faecal and saliva samples before cancer treatment. The investigators will also assess if there are any potential links between host microbial flora and chemoradiotherapy response

Study design:

Patients with a biopsy proven rectal adenocarcinoma have staging investigations, and these are discussed at a Colorectal Cancer (CRC) Multi- Disciplinary Team (MDT). If the CRM is threatened or involved then it would be standard practice to recommend pre-operative radiotherapy.

The 1st step for eligible patients is allocation to a consultant colorectal surgeon, who will meet the patient to confirm the standard plan for treatment.

The 2nd step is arranging an out-patient appointment to see a clinical oncologist. At this appointment the rationale, practical aspects and potential side effects of pre-operative therapy are discussed. In addition, the 3rd step, which is a discussion around the study plan, to collect and analyse both oral & faecal microbiota pre-pelvic treatment & again pre-surgery will be undertaken. A written patient information sheet is given to the patient to consider at home.

Pelvic radiotherapy is given as an out-patient. The first step is contouring the relevant anatomy, including tumour & associated lymph nodes, as well as normal organs that we want to limit the dose of radiation received. This contouring & preparation of a radiotherapy plan can take up to two weeks, so there is plenty of time for the 4th step, namely the patient considering whether they wish to take part in the study. If the patient decides to enter the study, they will sign & date a consent form.

Step 5 - For patients who decide to enter the study, the 5th step is arranging for collection of both oral & faecal samples for analysis before starting the pelvic radiotherapy (as an out-patient). The oral sample will be collected in the radiotherapy department prior to the first treatment, and the patient can choose to collect the faecal sample either at home or in the clinic, both on the day they are due to start the radiotherapy.

The patient continues on the radiotherapy and on completion there is a deliberately a 7 to 8 week wait, to allow the treatment to have an effect on the tumour, as well as allowing for any side effects to settle. After the treatment gap, the patient has another pelvic MRI scan, reviewed at a CRC MDT, to assess if the CRM is now clear, allowing the patient to proceed to potentially curative surgery.

Step 6 - For patients with a clear CRM a second set of oral & faecal samples for analysis will be collected the day prior to surgery. Again the patient has the option of collecting the faecal donation at home, and bringing it with them, or in clinic.

Step 7 - The surgical specimen is collected from theatre & brought directly to the pathology department by a member of the biodepository staff, as per standard practice. The pathologist, together with a member of the biodepository staff will collect samples from the lumen of the specimen, from the tumour & distant normal mucosa for microbiota & metabolite analysis. The tumour itself is assessed using a standardised approach, and any response graded using a validated & published system.

Step 8 - Comparison of the results pre- post- pelvic radiotherapy microbiota & metabolites, and an initial comparison with the pathology response grading. As there is a 15-20% possibility of a complete clinical response (cCR), these patients may wish to enter the 'active surveillance' programme. The faecal and oral microbiota of the cCR will also be analysed during this study. The samples of those individuals who do not have a clear CRM and do not progress to surgery will be analysed as a separate subgroup of the cohort

There will be no requirement for additional clinic visits for any patients taking part in the study. There will be additional time during the initial clinic visits, to discuss the study & answer any questions. Obtaining written consent will be timed with one of the visits for radiotherapy planning & preparation, and, as there is a 60 minute wait for oral contrast to reach the small bowel during the first radiotherapy CT simulator visit, there will not be any additional time waiting for the patient.

The collection of all study samples will be coordinated with routine visits to hospital, to ensure no additional visits would be required for a patient taking part in the study. A total of 25 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a locally advanced rectal cancer (defined as CRM threatening on MRI scans) in whom neoadjuvant chemoradiotherapy has been offered before consideration of curative resection
* must be able to consent to inclusion in project

Exclusion Criteria:

* Anyone who does not consent for inclusion
* Any non rectal adenocarcinoma
* Early rectal cancers that do not require neoadjuvant therapy
* Patients presenting as an emergency with an obstructing rectal cancer requiring an early resection
* Patients who are treated with short course radiotherapy alone rather than long course chemoradiotherapy

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Locally advanced rectal cancer patients suitable for neoadjuvant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
16s rRNA pyrosequencing analysis of microbial flora of rectal cancer patients | 1 year
  The microbial flora of the saliva and faeces of patients will be analysed at two time points. 1. before neoadjuvant chemoradiotherapy and 2. prior to surgery. This will be 16SrRNA pyrosequencing analysis to plot the microbial flora of each sample

SECONDARY OUTCOMES:
Categorisation of microbial flora against response to neoadjuvant chemoradiotherapy | 1 year
  The pathology resection specimen will be divided into four categories in terms of response to neoadjuvant chemoradiotherapy. 1. complete response, 2. good partial, 3, minimal and 4. complete response. These groupings will be used to analyse if there are any differences in microbial flora which may be able to predict for response to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided